CLINICAL TRIAL: NCT02724605
Title: Is Intraoperative Red Blood Cells Transfusion With Different Storage Duration Has Effect on Some Biochemical Parameters in Pediatric Trauma Patients Need Intraoperative Transfusion?
Brief Title: The Effect of Red Blood Cells Storage Duration on Biochemical Changes in Pediatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abdelrady S Ibrahim, MD (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Abdelrady S Ibrahim, MD, Assistant professor of Anesthesia and Intensive care, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB0000871236
Record Dates: First submitted 2016-03-20; First posted 2016-03-31 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Red Blood Cells Transfusion
Keywords: RBCS,; Transfusion,; Pediatric; Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): Red blood cells unit age 14 days or less
  Interventions: Biological: Red blood cells unit age 14 days or less
- Group B (Other): Red blood cells unit age more than 14 days
  Interventions: Biological: Red blood cells unit age more than 14 days

INTERVENTIONS:
Biological: Red blood cells unit age 14 days or less — 30 Patients who will receive units of packed red blood cells stored stored for 14 days or less
  Arms: Group A
Biological: Red blood cells unit age more than 14 days — 30 patients who will receive units of packed red blood cells stored for more than 14 days
  Arms: Group B

SUMMARY:
The aim of the study is to detect if the storage duration of red blood cells has impact on some biochemical parameters after intra operative transfusion in pediatric trauma patient

DETAILED DESCRIPTION:
* A pretransfusion draw of a few drops of patient venous blood, send for analysis by i-STAT Portable Clinical Analyser. Samples are processed immediately and provide laboratory quality results in 2 minutes using the CHEM 8+ i-STAT cartridge for measurement of:

  1. Potassium (K)
  2. Ionized Calcium (iCa)
  3. Glucose (Glu)
  4. Urea Nitrogen (BUN)/Urea
  5. Hemoglobin (Hb) and Hematocrit (Hct).
* Concurrently, a few drops of blood will be taken from the unit to be transfused will be analysed by i-STAT Portable Clinical Analyser for measurement of previous biochemical parameters.
* The details of the unit, such as draw date, volume of transfusion, and date of transfusion, will be recorded. The RBC unit will be delivered to the operative room from the blood bank in an insulated box.
* The transfusion is then given as clinically indicated at a rate of 50 to 150 mL/h based on the clinician's orders, the patient's weight, and the patient's clinical situation.
* Volumes will be transfused to children according to the following top-up transfusion equation: desired Hemoglobin (Hb) (g/dl) - actual Hemoglobin (Hb) (g/dl) x weight (kg) x 3. (usually 10-20 ml/kg).
* A second patient blood sample will be drawn one hour after the transfusion and will be analyzed by i-STAT Portable Clinical Analyser.
* Patient information will be recorded for age, weight, sex, and primary diagnosis.
* Demographic and clinical variables will be collected, to include type and quantity of all blood products and fluids received and medications administered. All surgical procedures will be documented.

ELIGIBILITY:
Inclusion Criteria:

.ASA I-II physical status patients.

* Genders Eligible for Study : both .
* Age: 2_10 years
* All non-crush trauma pediatric patients need intraoperative RBC transfusion.
* RBCs transfusion Volume within 10-20ml/kg.

Exclusion Criteria:

* Patients with renal failure (serum creatinine 1.5 mg/dL)
* Hepatic insufficiency.
* Furosemide diuresis.
* Succinylcholine for rapid sequence induction.
* Electrolytes disorders.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Serum potassium level | One hour after red blood cells transfusion
  Mmol/l

SECONDARY OUTCOMES:
Serum ionised calcium | One hour after red blood cells transfusion
  mg/dl
Serum glucose level | One hour after red blood cells transfusion
  Mmol/l
Blood Urea Nitrogen | One hour after red blood cells transfusion
  mg/dL
Hemoglobin level | One hour after red blood cells transfusion
  g/dl

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady S Ibrahim, Principal Investigator — Assistant professor of anesthesia and intensive care
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qu L, Triulzi DJ. Clinical effects of red blood cell storage. Cancer Control. 2015 Jan;22(1):26-37. doi: 10.1177/107327481502200105. PMID 25504276